CLINICAL TRIAL: NCT04889586
Title: Hand Motor Recovery Using a EMG-biofeedback in Stroke Rehabilitation: a Cross-sectional Study
Brief Title: Hand MOtor Rehabilitation Using a EMG-biofeedback: a Cross-sectional Study
Acronym: MORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Responsible Party: Principal Investigator, Andrea Turolla, Laboratory of Rehabilitation Technologies, IRCCS San Camillo, Venezia, Italy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2016.29
Record Dates: First submitted 2021-05-06; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Stroke; Stroke Hemorrhagic; Stroke, Ischemic; Hemiparesis; Hemiplegia
Keywords: Neurological Rehabilitation; Upper Extremity; Electromyography; Hand Gesture
MeSH Terms: conditions — Stroke; Hemorrhagic Stroke; Ischemic Stroke; Paresis; Hemiplegia

STUDY DESIGN:
Intervention Model Description: Each subject is assessed with a clinical protocol and an instrumental test, consists in executing 10 hand gestures by wearing a EMG-biofeedback armband
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): The subjects were clinically assessed with a define clinical protocol. After that, the subjects executed the device test with EMG-biofeedback wearable armband.
  Interventions: Device: EMG-biofeedback armband (REMO)

INTERVENTIONS:
Device: EMG-biofeedback armband (REMO) — After clinical evaluation, the subjects execute an instrumental test. By wearing EMG-biofeedback device (REMO), the subjects have to perform 10 different hand gestures: thumb abduction, pinch, finger flexion, finger extension, wrist flexion, wrist extension, forearm pronation, forearm supination, radial wrist deviation and ulnar wrist deviation. The muscle activations (EMG signals) during the execution of each movements, are recorded for 3 seconds.

SUMMARY:
Recovery of upper limb and hand gestures is fundamental for autonomy restoration after stroke. Innovative technologies are a valid support for the delivery of rehabilitation treatments. Embedding surface electromyographic (sEMG) into wearable devices, allows the customisation of rehabilitation exercises, based on the clinical profile of each patient.

DETAILED DESCRIPTION:
The aims of this study are to determine safety and feasibility of a prototype EMG-control wearable device (REMO) and to individualise clinical features of stroke survivors able to control the EMG armband targeted to hand rehabilitation.

The device REMO consists in an armband composed by 8 bipolar electrodes able to record and process the electromyography of forearm muscles. The patterns of muscle activations are classified and used to perform EMG-biofeedback exercises in stroke rehabilitation training. The device is developed by clinicians of IRCCS San Camillo Hospital and spin-off Morecognition Srl.

A total of 100 stroke patients patients has been recruited. They are clinically assessed and then tested on the ability to control the sEMG wearable device. The test is composed of 10 hand and fingers gestures to be performed with the paretic hand. Baseline and activation sEMG signals are recorded and compared for each movement. Three conditions representing absent, partial or full control of the device are defined and logistic multivarialbes regression models are used to identify clinical features describing the group each patient belongs to. Clinical cut-off for each strata is identified by odds ratio.

ELIGIBILITY:
Inclusion Criteria:

* Single ischemic or haemorrhagic stroke;
* Score lower than 100 out of a total of 126 at the Functional Independence Measure (FIM) scale

Exclusion Criteria:

* Untreated epilepsy;
* Major depressive disorder;
* Fractures;
* Traumatic Brain Injurj;
* Severe Ideomotor Apraxia;
* Severe Neglect;
* Severe impairment of verbal comprehension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2019-02-11 (Actual); Study Completion 2019-02-27 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Upper Extremity (FMA-UE) | within 1 week from enrolment.
  Motor function of the upper limb is measured by means of the Fugl-Meyer Scale. There are 3 values: 0 (severe impairment), 1 (moderate impairiment), 2 (preserved function)

SECONDARY OUTCOMES:
Fugl-Meyer - sensation | within 1 week from enrolment.
  Sensation of the hemiparetic side is measured by means of the Fugl-Meyer Scale. There are 3 values: 0 (severe impairment), 1 (moderate impairiment), 2 (preserved function)
Fugl-Meyer - pain and Range of Motion | within 1 week from enrolment.
  Pain and Range of Motion of the hemiparetic upper limb is measured by means of the Fugl-Meyer Scale. There are 3 values: 0 (severe impairment), 1 (moderate impairiment), 2 (preserved function)
Box and Blocks Test (BBT) | within 1 week from enrolment.
  The patient has to carry as much cubes as possible, one by one, from a container to another one in one minute. The test is performed with both hands.
Reaching Performance Scale (RPS) | within 1 week from enrolment.
  RPS assesses the ability of subjects to reach an object (a cone). The cone is placed at both 4-cm (close) and 30-cm (far) distance from the subject. The subject is asked to reach and grab the cone if possible. The observer evaluates the quality of reaching instead of the grip strength (Total score = 36 points).
Modified Ashworth Scale (MAS) | within 1 week from enrolment.
  Spasticity is measured using the MAS of five muscles: Pectoralis major, biceps, wrist flexors, flexor digitorum superficialis, flexor digitorum profundus (Total score = 20 points).
Nine Hole Pegboard Test (NHPT) | within 1 week from enrolment.
  NHPT measures the dexterity of the hand. Patient should insert 9 pins in the board. There are 9 pins. The number of pins inserted in 50 sec are registered or if the patient inserted 9 pins, then the time is registered.
Functional Independence Measure scale (FIM) | within 1 week from enrolment.
  FIM is an 18-item scale that assesses the degree of autonomy in carrying out activities of daily living (total score = 126 points).
Number of movements controlled by EMG-biofeedback device | within 1 week from enrolment.
  The patient is able to control a movement with the device if he crosses the pre-defined empirical threshold (10%) of the ratio between the maximum voluntary contraction (MVC) of the movement and the EMG recording during baseline (i.e. rest position).

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Turolla, PhD, Principal Investigator — IRCCS San Camillo Hospital
Locations (1):
- IRCCS San Camillo Hospital, Venice-Lido, Venice, Italy

REFERENCES:
- [Background] Celadon N, Dosen S, Binder I, Ariano P, Farina D. Proportional estimation of finger movements from high-density surface electromyography. J Neuroeng Rehabil. 2016 Aug 4;13(1):73. doi: 10.1186/s12984-016-0172-3. PMID 27488270
- [Background] Dipietro L, Ferraro M, Palazzolo JJ, Krebs HI, Volpe BT, Hogan N. Customized interactive robotic treatment for stroke: EMG-triggered therapy. IEEE Trans Neural Syst Rehabil Eng. 2005 Sep;13(3):325-34. doi: 10.1109/TNSRE.2005.850423. PMID 16200756
- [Background] Paleari M, Di Girolamo M, Celadon N, Favetto A, Ariano P. On optimal electrode configuration to estimate hand movements from forearm surface electromyography. Annu Int Conf IEEE Eng Med Biol Soc. 2015;2015:6086-9. doi: 10.1109/EMBC.2015.7319780. PMID 26737680
- [Background] Pollock A, Farmer SE, Brady MC, Langhorne P, Mead GE, Mehrholz J, van Wijck F. Interventions for improving upper limb function after stroke. Cochrane Database Syst Rev. 2014 Nov 12;2014(11):CD010820. doi: 10.1002/14651858.CD010820.pub2. PMID 25387001